CLINICAL TRIAL: NCT06864871
Title: Complications in Minimally Invasive Aesthetic Dermatological Procedures in Switzerland: A Descriptive Study From a University Referral Center
Brief Title: Complications in Minimally Invasive Aesthetic Dermatological Procedures in Switzerland
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00297; th25Vasconcelos
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Aesthetic Procedures; Complication of Treatment
Keywords: Minimally Invasive Procedures; Injectable Procedures; Non-injectable Procedures; Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this retrospective study is to describe cases of complications from minimally invasive aesthetic procedures treated at a university reference centre in Switzerland between 2021 and 2024.

DETAILED DESCRIPTION:
During the past decade, a steady increase in aesthetic procedures has been observed. Over the last four years, non-surgical procedures have grown by 40%. The five most popular treatments are botulinum toxin, hyaluronic acid, hair removal, chemical peels, and nonsurgical fat reduction.

With the increase in aesthetic procedures, adverse effects have also increased. Contributing factors include weak regulations, unlicensed practice, and individuals with little or no formal training administering botulinum toxins and dermal fillers.

This study aims to analyze unexpected and often unfavorable outcomes, referred to as complications, arising from minimally invasive procedures-both non-injectable (e.g., laser treatments, chemical peels) and injectable (e.g., botulinum toxin, fillers). The complications are categorized based on their severity and ethiology. This retrospective case series is conducted at a university reference center in Switzerland (Margarethenklinik of the University Hospital Basel) between January 2021 and December 2024.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older of all genders, ethnic and social demographic background that have signed the General consent and the Photo-Informed Consent Form.

Exclusion Criteria:

* Patients who didn't sign the general consent.
* Patients under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that had an appointment at Margarethenklinik of the University Hospital Basel between January 2021 and December 2024.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Total cases of complications | Between January 2021 and December 2024
  The total number of complications from minimally invasive aesthetic procedures treated at a university reference centre in Switzerland between 2021 and 2024 is analyzed and classified by ethiology and severity.
Type of aesthetic procedure | Between January 2021 and December 2024
  The type of aesthetic procedure that led to the complication is analyzed and classified by ethiology and severity.
Diagnosis of complication | Between January 2021 and December 2024
  The diagnosis of complication is analyzed and classified by ethiology and severity.

SECONDARY OUTCOMES:
Location of aesthetic procedure (Switzerland or abroad) | Between January 2021 and December 2024
  The location where the aesthetic procedure was performed is analyzed, whether in Switzerland or abroad. For procedures conducted in Switzerland, the specific canton where the treatment took place will be documented.
Type of practitioner performing the aesthetic procedure | Between January 2021 and December 2024
  The type of practitioner who has performed the aesthetic procedure is analyzed, whether it was by a physician, another authorized professional, or an unlicensed practitioner.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Vasconcelos Berg, MD, PhD, Principal Investigator — Margarethenklinik, University Hospital Basel
Locations (1):
- Margarethenklinik, University Hospital Basel, Basel, Switzerland